CLINICAL TRIAL: NCT00108381
Title: Efficacy of Tailored Cognitive-Behavioral Therapy for Chronic Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: MHBS042-03
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Back Pain
Keywords: chronic back pain; cognitive-behavioral; pain; stages of change
MeSH Terms: conditions — Back Pain; Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Standard and Tailored Conditions
  Interventions: Behavioral: tailored cognitive behavior therapy; Behavioral: standard care

INTERVENTIONS:
Behavioral: tailored cognitive behavior therapy — tailored psychological treatment
Behavioral: standard care — standard psychological treatment

SUMMARY:
This clinical trial compares two psychological treatments for back pain.

DETAILED DESCRIPTION:
The primary objective is to examine the incremental efficacy of a patient-centered and tailored self-management treatment approach, Tailored Cognitive-Behavior Therapy (TCBT), for persons with chronic musculoskeletal pain. TCBT will be compared with a Standard Cognitive- Behavior Therapy (SCBT) condition. The hypothesis is that TCBT will be associated with improved outcomes following treatment. Outcome will be assessed by multiple standardized measures of key domains of the chronic pain experience. Secondary objectives are to examine the process of successful self-management treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic back pain for at least 6 months
* Treatment by medication or physical therapy

Exclusion Criteria:

* Acute or life threatening physical illness
* Current alcohol or substance abuse or dependence
* Current psychosis or suicidal ideation treatment by anesthesiology, chiropractic care or surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2004-01; Primary Completion 2010-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Multiple standardized measures of key domains of the chronic pain experience | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Kerns, PhD, Principal Investigator — VA Connecticut Health Care System (West Haven)
Locations (1):
- VA Connecticut Health Care System (West Haven), West Haven, Connecticut, United States

REFERENCES:
- [Result] Finan PH, Burns JW, Jensen MP, Nielson WR, Kerns RD. Pain coping but not readiness to change is associated with pretreatment pain-related functioning. Clin J Pain. 2012 Oct;28(8):687-92. doi: 10.1097/AJP.0b013e3182400867. PMID 22688600
- [Result] Kerns RD, Burns JW, Shulman M, Jensen MP, Nielson WR, Czlapinski R, Dallas MI, Chatkoff D, Sellinger J, Heapy A, Rosenberger P. Can we improve cognitive-behavioral therapy for chronic back pain treatment engagement and adherence? A controlled trial of tailored versus standard therapy. Health Psychol. 2014 Sep;33(9):938-47. doi: 10.1037/a0034406. Epub 2013 Dec 2. PMID 24295024
- [Derived] Burns JW, Nielson WR, Jensen MP, Heapy A, Czlapinski R, Kerns RD. Does Change Occur for the Reasons We Think It Does? A Test of Specific Therapeutic Operations During Cognitive-Behavioral Treatment of Chronic Pain. Clin J Pain. 2015 Jul;31(7):603-11. doi: 10.1097/AJP.0000000000000141. PMID 25119513
- [Derived] Burns JW, Nielson WR, Jensen MP, Heapy A, Czlapinski R, Kerns RD. Specific and general therapeutic mechanisms in cognitive behavioral treatment of chronic pain. J Consult Clin Psychol. 2015 Feb;83(1):1-11. doi: 10.1037/a0037208. Epub 2014 Jun 30. PMID 24979313